CLINICAL TRIAL: NCT03371537
Title: Study of Hemodynamic Conditions Measured During Hepatectomy
Acronym: DEBIFOIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/DEBIFOIE; 2017-A01754-49 (Other: IdRCB); 2017-61 (Other: CPP)
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Liver Dysfunction; Circulatory; Change
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatectomy: Patient undergoing laparotomy for liver resection. The aim is to measure the flow rates in the portal vein and the hepatic artery.
  Interventions: Procedure: Liver debit measure

INTERVENTIONS:
Procedure: Liver debit measure — Mesure of liver debit during hepatectomy

SUMMARY:
Hepatocellular insufficiency is a dreaded complication after hepatectomy, since, if it is persistent, it leads to the death of the patient in the absence of liver transplantation.

The preoperative evaluation aims in particular to estimate the risk of postoperative hepatocellular insufficiency so as to minimize or contraindicate high-risk patients.

It has been shown that the flow of the portal vein is correlated with liver function, especially in the living donor and after portal embolization. More recently, the study of flow rates in the portal vein and the hepatic artery after transplantation has shown a correlation with the recovery of graft function.

The hypothesis is that portal and arterial flow after hepatectomy can predict postoperative hepatocellular function.

DETAILED DESCRIPTION:
Measurements of flow rates in the portal vein and the hepatic artery by different transit times are available thanks to the Medistim VeriQTM system that the investigators already use routinely in the context of liver transplantation when performing hepatectomies.

ELIGIBILITY:
Inclusion Criteria:

* patient 18 years or more
* Patient undergoing laparotomy for liver resection

Exclusion Criteria:

* Patient under tutorship or curatorship
* Pregnant or lactating woman
* Difficulties in understanding French
* Patient operated by laparoscopy
* Patient having objected to the processing of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing laparotomy for liver resection
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Liver vessel debit | Baseline
  Mesure of liver debit during hepatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ephrem SALAME, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Service de Chirurgie Digestive, Oncologique, Endocrinienne et Transplantation Hépatique, CHRU de TOURS, Tours, France